CLINICAL TRIAL: NCT05846230
Title: A Randomised, Double-blind, Parallel Group, Roll-over Study Evaluating Long-term Safety and Efficacy of Oral Doses of BI 1291583 q.d. in Patients With Bronchiectasis (Clairleafᵀᴹ)
Brief Title: Clairleafᵀᴹ: A Study to Test Long-term Treatment With BI 1291583 in People With Bronchiectasis Who Took Part in a Previous Study With This Medicine
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1397-0017; 2023-503290-38-00 (Registry Identifier: CTIS); U1111-1292-0921 (Registry Identifier: WHO Registry)
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BI 1291583 low dose arm (Experimental)
  Interventions: Drug: BI 1291583; Drug: Placebo matching BI 1291583
- BI 1291583 medium dose arm (Experimental)
  Interventions: Drug: BI 1291583; Drug: Placebo matching BI 1291583
- BI 1291583 high dose arm (Experimental)
  Interventions: Drug: BI 1291583; Drug: Placebo matching BI 1291583

INTERVENTIONS:
Drug: BI 1291583 — Tablet
  Other Names: Verducatib
Drug: Placebo matching BI 1291583 — Tablet

SUMMARY:
This study is open to adults aged 18 years and older with bronchiectasis. People can join the study if they were previously enrolled in another study with BI 1291583 (1397-0012: Airleafᵀᴹ or 1397-0013 Clairaflyᵀᴹ). The purpose of this study is to find out whether a medicine called BI 1291583 helps people with bronchiectasis, an inflammatory lung condition. The investigators also want to know how well people with this condition can tolerate BI 1291583 in the long term.

Participants take a low, medium, or high dose of BI 1291583 as a tablet once a day for up to 1 year. Participants who were taking placebo in the AirleafTM or ClairaflyTM study are put into the BI 1291583 dosage groups randomly, which means by chance. Placebo tablets look like BI1291583 but do not contain any medicine. Participants who were taking BI 1291583 in the AirleafTM or ClairaflyTM study continue to take the same dose.

Participants visit the study site 10 times and get 4 phone calls from the site staff. During the visits, the doctors collect information on any health problems of the participants. The doctors also check whether BI 1291583 helps reduce the symptoms of bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the treatment period in Phase II trials (1397-0012 or 1397-0013) as planned per protocol.
* Male or female patients. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly, as well as one barrier method. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent prior to admission to the trial, in accordance with Good Clinical Practice (GCP) and local legislation.

Exclusion Criteria:

Laboratory and medical examination

* Moderate or severe liver disease (defined by Child-Pugh score B or C hepatic impairment) or aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3.0x Upper limit of normal (ULN) at Visit 1 (or at the last safety assessment in the parent trial, if no more than 6 weeks passed since then).
* Estimated glomerular filtration rate (eGFR) according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula <30 mL/min at Visit 1 (or at the last safety assessment in the parent trial, if no more than 6 weeks passed since then).
* An absolute blood neutrophil count <1,000/mm^3 (equivalent to <1,000 cells/μL or <10^9 cells/L) at Visit 1 (or at the last safety assessment in the parent trial, if no more than 6 weeks passed since then).
* Any findings in the medical examination and/or laboratory value assessed at Visit 1 (or at the last safety assessment in the parent trial, concerning the lab tests, if no more than 6 weeks passed since then), that in the opinion of the investigator may put the patient at risk by participating in the trial.

New concomitant diagnosis and therapy

* A new diagnosis of

  * Hypogammaglobulinemia
  * Common variable immunodeficiency
  * α1-antitrypsin deficiency being treated augmentation therapy
  * Allergic bronchopulmonary aspergillosis being treated or requiring treatment
  * Tuberculosis or non-tuberculous mycobacterial infection being treated or requiring treatment according to local guidelines
  * Palmoplantar keratosis; or keratoderma climactericum
  * Hypothyroidism, myxedema, chronic lymphedema with associated hyperkeratosis of the skin, acrocyanosis. If a subject has hypothyroidism but is treated and compensated, the subject is allowed into the trial
  * Psoriasis affecting palms and soles; or body surface area for psoriasis ≥10%
  * Reactive arthritis (Reiter's syndrome); keratoderma blennorrhagicum
  * Pityriasis rubra pilaris
  * Atopic dermatitis affecting palms and soles; or body surface area for atopic dermatitis ≥10%
  * Active extensive verruca vulgaris, as per investigator's discretion
  * Active fungal infection of hand and/or feet not adequately treated and responsive to antifungal therapy, as per investigator's discretion.
* Any clinically relevant respiratory infection within 4 weeks prior Visit 2, unless recovered in the opinion of the investigator by Visit 2.
* Any acute infection requiring systemic or inhaled anti-infective therapy within 4 weeks prior Visit 2.
* Positive serological tests for hepatitis B, hepatitis C (also confirmed with ( Hepatitis C Virus ribonucleic acid test (HCV RNA))), or human immunodeficiency virus (HIV) infection, or known infection status at Visit 2. (The test results will be available after randomisation. In case the results no longer satisfy the entry criteria, these patients will be discontinued.)
* Any new evidence of a concomitant disease, such as Papillon-Lefèvre Syndrome (PLS), relevant pulmonary, gastrointestinal, hepatic, renal, cardiovascular, metabolic, immunological, hormonal disorders, or patients who are immunocompromised with a higher risk of invasive pneumococcal disease or other invasive opportunistic infections (such as histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis), that in the opinion of the investigator, may put the patient at risk by participating in the trial.
* Received any live attenuated vaccine within 4 weeks prior to Visit 1.
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse events (TEAEs) | up to 12 months

SECONDARY OUTCOMES:
Time to first pulmonary exacerbation from first drug administration in this trial to the end of the trial | up to 12 months
  A pulmonary exacerbation in this trial is defined as having three or more of the following symptoms for at least 48 hours resulting in a physician's decision to prescribe antibiotics (oral or intravenous):
  * Increased cough
  * Increased sputum volume or change in sputum consistency
  * Increased sputum purulence
  * Increased breathlessness and/or decreased exercise tolerance
  * Fatigue and/or malaise
  * Hemoptysis
Rate of pulmonary exacerbations (number of events per person-time) over the course of this trial | up to 12 months

CONTACTS AND LOCATIONS:
Locations (102):
- United States (11):
  - Newport Native MD, Inc, Newport Beach, California
  - University of California Davis, Sacramento, California
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - New York University Langone Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Metroplex Pulmonary & Sleep Center, McKinney, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
- Australia (6):
  - Macquarie University, Macquarie Park, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Lung Research Queensland, Chermside, Queensland
  - Mater Research Institute, South Brisbane, Queensland
  - Institute for Respiratory Health, Nedlands, Western Australia
  - Trialswest, Spearwood, Western Australia
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Bulgaria (5):
  - Medical Center "Zdrave-1", Kozloduy
  - Medica Center Hera - Montana Branch, Montana
  - Medical Center ReSpiro Ltd, Razgrad
  - SHATPPD "Dr. Dimitar Gramatikov", Rousse
  - Medical Center Hera EOOD, Sofia
- Canada (2):
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Czechia (2):
  - Pulmonary Private Practice Kralupy, Kralupy nad Vltavou
  - The First Pulmonary Private Practice, Prague
- Denmark (6):
  - Aalborg Sygehus Syd, Aalborg
  - Hvidovre Hospital, Hvidovre
  - Copenhagen University Hospital, Rigshospitalet, København Ø
  - Odense University Hospital, Odense
  - Sjællands Universitetshospital, Roskilde
  - Vejle University Hospital, Vejle
- France (3):
  - CHU Amiens-Picardie, Amiens
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pontchaillou, Rennes
- Germany (11):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - IKF Pneumologie GmbH & Co. KG, Frankfurt
  - Velocity Clinical Research Germany GmbH, Ahrensburg, Großhansdorf
  - Medizinische Hochschule Hannover, Hanover
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitätsklinikum Jena, Jena
  - Klinikum Konstanz, Konstanz
  - Velocity Clinical Research Germany GmbH, Lübeck, Lübeck
  - Klinikum der Universität München AÖR, München
  - Velocity Clinical Research Germany GmbH, Wiesbaden, Wiesbaden
- Hungary (2):
  - Semmelweis University, Budapest
  - Da Vinci Private Clinic, Pécs
- Israel (4):
  - Soroka Univ. Medical Center, Beersheba
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Meyer, Florence
  - Policlinico "Paolo Giaccone", Palermo
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (11):
  - Nagoya University Hospital, Aichi, Nagoya
  - Hirosaki University Hospital, Aomori, Hirosaki
  - Kameda Clinic, Chiba, Kamogawa
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Ibarakihigashi National Hospial, Ibaraki, Naka-gun
  - Kagoshima University Hospital, Kagoshima, Kagoshima
  - Matsusaka City Hospital, Mie, Matsusaka
  - Osaka Toneyama Medical Center, Osaka, Toyonaka
  - Saga University Hospital, Saga, Saga
  - Fukujuji Hospital, Tokyo, Kiyose
  - Kitasato Institute Hospital, Tokyo, Minato-ku
- Latvia (6):
  - Med.Center OLVI Health Center Assotiation,Private Practice, Daugavpils
  - Daugavpils Regional Hospital LTD Centre Outpatient Clinic, Daugavpils
  - VCA Dubultu Medical center, Jūrmala
  - Riga 1st Hospital, Riga
  - Pauls Stradins Clinical University Hospital, Riga
  - LUMPII Doctors practice, Riga
- Mexico (5):
  - Mediadvance Clinical S.A.P.I de C.V., Chihuahua City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Hospital Universitario Nuevo de Nuevo León - CEPREP, Monterrey, Nuevo León
  - Oaxaca Site Management Organization, S.C., Oaxaca City
  - Clinical Research Institute S.C., Tlalnepantla
- Netherlands (3):
  - Amsterdam UMC, location VUMC, Amsterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Gelre Ziekenhuis Zutphen, Zutphen
- Poland (5):
  - Respiratory Medicine Centre, private prac., Bialystok, Bialystok
  - Screenmed Sp. z o.o., Piaseczno
  - Alergopneuma Medical Center, Świdnik
  - Altamed Specjalistyczna Praktyka Lekarska Pawel Sliwinski, Warsaw
  - Dr. Piotr Napora, Center of Clinical Research, Wroclaw
- ULS de Santa Maria, E.P.E, Lisbon, Portugal
- South Korea (5):
  - Chungbuk National University Hospital, Cheongju-si
  - Asan Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
- Spain (5):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital de Mérida, Mérida
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
- Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul, Turkey (Türkiye)
- Ninewells Hospital & Medical School, Dundee, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Badorrek P, Diefenbach C, Kogler H, Eleftheraki A, Seitz F, Hohlfeld JM. Novel cathepsin C inhibitor, BI 1291583, intended for treatment of bronchiectasis: Phase I characterization in healthy volunteers. Clin Transl Sci. 2024 Aug;17(8):e13891. doi: 10.1111/cts.13891. PMID 39175217
- See also: Related Info — http://mystudywindow.com